CLINICAL TRIAL: NCT02300090
Title: A Real-World Assessment of a COPD Disease Management Support Service (Me & My COPD).
Acronym: Me&MyCOPD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 149902
Record Dates: First submitted 2014-11-21; First posted 2014-11-24 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, Exacerbation, respiratory disease, lung disease, breathlessness, dyspnoea, sputum, wheezing, cough
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiration Disorders; Lung Diseases; Dyspnea; Respiratory Sounds; Cough | interventions — Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention group: This group of patients (n=250) will receive the digital service (smart phone application and bluetooth inhaler device) in addition to current best care from their healthcare professional.
  Interventions: Device: Test Group
- Control group: This group of patients (n=250) will receive current best care alone. Control patients will not have access to the digital service.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Test Group — Patients receive a mobile phone with the Me & My COPD app installed. Patients also receive a bluetooth inhaler device that is fitted to their usual reliever inhaler.
  Groups: Intervention group
Other: Control Group — Patients in the control group receive only standard care; there are no interventions within this group of patients
  Groups: Control group

SUMMARY:
A real world study to determine the effectiveness of a patient support service to aid COPD patients in their self management.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate a digital health wellness support tool for patients in primary care with COPD using a smart mobile app, patient web portal and technology attached to the patients SABA reliever inhaler. Using the patients pre-defined COPD self management plan, the active arm of the study complete a daily diary (EXACT PRO) and record their daily SABA inhaler usage. After defining a health and symptom score baseline over a two week period, any significant deviations in SABA reliever use or daily diary scoring will alert patients that they may be having a change in their symptoms and advise them to refer to their self management plan and if they need to start their rescue medication. The primary outcome measure for the study is a 25% reduction in unplanned COPD hospital admissions (n=250 completing the study in each arm).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD
* FEV1/FVC ratio >0.3-<0.7 and FEV1 > 30% post-bronchodilator
* Prescribed either ICS, LABA and or LAMA at dose for COPD
* Exacerbations reported within the last 12 months requiring treatment with >1 systemic steroid and/or antibiotics, OR hospitalisation within last 12 months due to exacerbation, OR have received >12 SABA prescriptions in previous 12 months
* Patient has a self management plan which includes use of an oral steroid at a dose within NICE guidelines, and additionally antibiotics as appropriate.

Exclusion Criteria:

* Symptomatic asthma or seasonal allergic rhinitis leading to hospitalisation in previous 12 months
* Patients unable to use a mobile phone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and females, of any age with a clinical diagnosis of COPD
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
To detect a reduction in the rate of hospitalisations due to COPD exacerbations | Analysed over a twelve month timeframe
  The mean number of COPD related hospitalisations per patient per year for patients who are receiving the digital service in the study will be compared to the rate of COPD related hospitalisations in patients receiving current best care alone over a twelve period.

SECONDARY OUTCOMES:
To detect a reduction in the duration of hospitalisations due to COPD exacerbations. | 12 months
  The average duration of COPD related hopspitalisations (number of bed days) per patient will be compared across patients receiving the digital service and those receiving current best care alone.
To detect a reduction in the number of exacerbations requiring treament with antibiotics and or systemic steriods | 12 months
  The number of exacerbations requiring treament with antibiotics and or systemic steriods will be compared across patients receiving the digital service and those receiving current best care alone.
To detect an improvement in patients own perceived health status, as assessed by St Georges Respiratory Questionnaire-C | 12 months
  The patients assessment of their own health status will be assessed over time using the St Georges Respiratory Questionnaire-C, and will be compared across patients receiving the digital service and those receiving current best care alone.

OTHER OUTCOMES:
To detect a difference in the use/prescribing of maintenance therapy | 12 months
  To detect a difference in the use/prescribing of maintenance therapies (inhaled corticosteroids/long acting beta agonists and or long acting muscarinic antagonists) by comparison of repeat prescriptions across patients receiving the digital service and those receiving current best care alone.
To detect a difference in the use/prescribing of reliever therapy | 12 months
  To detect a difference in the use/prescribing of reliever therapy, as measured through repeat prescriptions, by comparison of patients receiving the digital service and those receiving current best care.
To assess patinet engagement in the use of the digital service | 12 months
  To assess the engagement of patients receiving the digital service as measured by frequency of access to infromational content and goal management.

CONTACTS AND LOCATIONS:
Overall Officials: David MG Halpin, MBBS, MRCP, FRCP, Principal Investigator — Royal Devon and Exeter Hospital
Locations (5):
- United Kingdom (5):
  - Research Site, East Cheshire, UK
  - Research Site, Liverpool, UK
  - Research Site, Manchester, UK
  - Research Site, Newcastle, UK
  - Research Site, Oldham, UK